CLINICAL TRIAL: NCT05178277
Title: Czech Alpha-1 Antitrypsin Deficiency Registry, the National Observational Study.
Brief Title: Czech AATD Registry
Status: Recruiting | Type: Observational
Sponsor: Thomayer University Hospital (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Jan Chlumsky, M.D., Principal Investigator, Thomayer University Hospital
Other Study IDs: IBA1115
Record Dates: First submitted 2021-11-12; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Alpha-1-antitrypsin Deficiency
Keywords: Alpha-1-antitrypsin deficiency; AATD; national registry
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Alpha-1-antitrypsin deficiency is the most common congenital disease of the respiratory system, leading to early pulmonary emphysema or bronchiectasis. Pulmonary involvement significantly accelerates active cigarette smoking. Patients with alpha-1-antitrypsin deficiency may also have liver cirrhosis, vasculitis, skin or intestinal disorders.

The AATD Registry is a non-interventional multicenter retrospective prospective longitudinal follow-up of patients with alpha-1-antitrypsin deficiency.

The aim of the AATD National Registry is to collect and analyze clinical data in patients with alpha-1 antitrypsin deficiency.

DETAILED DESCRIPTION:
Alpha-1 antitrypsin deficiency is a genetic disorder that may result in lung disease or liver disease. It is assume that it affects 1 person from a cohort of 2,000-5,000 people of the general population. Among patients with COPD, the incidence of the disorder is significantly higher. The prognosis of these patients is incomparably worse compared to classic COPD, because it affects younger patients and the rate of lung tissue loss is faster. The diagnosis is made in patients with pre-existing COPD by examination of the plasma concentration of AAT. In case of its reduction, genetic examination is added. The progression of the disease is rapid and has been shown to be slowed by lifelong augmentation treatment with human AAT. However, in routine clinical practice, it is very difficult to assess the effectiveness of treatment, the progression of lung disease or the prognosis of the disease.

The AATD registry is a non-interventional multicenter retrospective prospective longitudinal follow-up of patients with alpha-1-antitrypsin deficiency. The national registry collects data from all patients with severe or rare AAT deficiency, regardless of the type of organ impairment and age, and thus provides a view of this genetic variation in the Czech population.

The aim of the AATD Registry is to collect and analyse clinical data of patients with alpha-1 antitrypsin deficiency and increase the professional awareness of this hereditary disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with alpha-1-antitrypsin deficiency

Exclusion Criteria:

* Patient disagreement with inclusion in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with alpha-1-antitrypsin deficiency
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of lung function parameters over time | within one year after completion
  assessement of the rate of decline of FEV1 (ml, %predicted), measured annually
Changes of exercise tolerance tolerance over time | within one year after completion
  assessment of changes of peak oxygen consumption (peakVO2, ml/kg/min) measured every two years
Changes of respiratory function over time | within one year after completion
  assessement of the rate of decline of TLco (mol/min/kPa, %predicted), measured annually
Changes of quality of life over time | within one year after completion
  assessement of the rate of decline of COPD assessment test (CAT, points), measured annually
Relationship of pulmonary function and lung CT densitometry to better determine phenotypes of COPD due to AAT deficiency | within one year after completion
  Assessement of any possible relationship of primary outcomes 1-3 using LAA (low attenuation area, %) and distribution of emphysema (craniocaudal distribution of emhysema, points)

SECONDARY OUTCOMES:
Behavior of individuals with no or minimal lung involvement | within one year after completion
  Assessement of prognosis of deficient non-smokers by monitoring primary outcome parameters 1-3
Progression of other organ disorders, namely liver | within one year after completion
  Laboratory detection of changes in liver tests (ALT, AST, ALP, GGT, ukat/l)

CONTACTS AND LOCATIONS:
Overall Officials: Jan MD Chlumsky, PhD, Principal Investigator — Thomayer University Hospital
Locations (1):
- Thomayer university hospital, Prague, Czech Republic, Czechia